CLINICAL TRIAL: NCT03440632
Title: Functional Electrical Stimulation of the Ankle Dorsiflexors During Walking in Children With Unilateral Spastic Cerebral Palsy: a Randomized Crossover Intervention Study
Brief Title: Functional Electrical Stimulation During Walking in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL63250.068.17
Record Dates: First submitted 2017-11-20; First posted 2018-02-22 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy; Spastic; Foot Drop
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Peroneal Neuropathies

STUDY DESIGN:
Intervention Model Description: randomisation for the order of treatments and thereby for the total length of the 'conventional therapy phase'.
Who Masked: Outcomes Assessor
Masking Description: The physical examination and the advanced analysis of the 3D gait analysis will be done be a blinded examiner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FES start (Other): Start: 4 weeks 'adaptation phase' and 8 weeks 'FES phase'. Adaption phase: the stimulus (in Volt) will gradually be increased up to an effective level and the wear time has to be increased from 30 minutes to 6 hours a day. FES phase: the participants have to wear the FES device for minimal 6 hours a day during walking. Usual physiotherapy can be continued during the FES phase.
  Second: after the FES phase, this group will enter the 'wash-out' period of 6 weeks for fading of the therapeutic effects, in which they return to their conventional therapy. Afterwards, 12 weeks of conventional therapy (orthoses/shoes and usual physiotherapy) with measurements at start and end will follow.
  Interventions: Device: FES
- Conventional start (Other): Start: wearing usual orthoses/shoes on a daily basis for the first 12 weeks of the study. Usual physiotherapy can be continued.
  Second: after 12 weeks this group will enter a 6 week watch out phase, and next be switched to FES treatment for 12 weeks, consisting of: 4 weeks 'adaptation phase' with gradual increase of the treatment and 8 weeks 'FES phase'.
  Interventions: Device: FES

INTERVENTIONS:
Device: FES — Functional electrical stimulation of the ankle dorsiflexors during walking, using a (superficial) neurostimulator with tilt sensor.

SUMMARY:
Children with spastic cerebral palsy (CP) often walk with insufficient ankle dorsiflexion in the swing phase. A pathological gait, known as drop-foot gait, can be the result and this has 2 major complications: foot-slap during loading response and toe-drag during swing. This is partly caused by weakness of the anterior tibial muscle and partly due to co-contraction of both the fibular- and anterior tibial muscle. For classification of gait, the Winters scale can be used, where unilateral CP with dropfoot is classified as type I.

In daily life these problems cause limited walking distance and frequent falls, leading to restrictions in participating in daily life. The current guideline for spastic cerebral palsy describes the following therapies: 1) conservative therapy (physiotherapy, orthopaedic shoes and orthoses) 2) drugs suppressing spasticity 3) surgical interventions.

Functional electrical stimulation (FES) may be an effective alternative treatment for children with spastic CP and a drop foot. By stimulating the fibular nerve or the anterior tibial muscle directly during the swing phase, dorsiflexion of the foot is stimulated. In contrast to bracing, FES does not restrict motion, but does produce muscle contraction, and thus has the potential to increase strength and motor control through repetitive neural stimulation over time.

In a systematic review the investigators found that FES immediately improves ankle dorsal flexion and reduces falls and these effects also sustain. However, it should be noted that the level of evidence is limited. Until now, the use of FES in CP is limited and no data exist about the effects on walking distance (activity level) and participation level.

The overall objective of this study is to conduct a randomised cross-over intervention trial in children with unilateral spastic CP with 12 weeks of FES (for every participant) and 18 weeks of conventional therapy. The effectiveness of FES will be examined at participation leven, using individual goal attainment. Next to that the effect at gait will be measured. An additional goal is to investigate the cost effectiveness of FES, which, in case of a positive effect, may support allowance by insurance companies.

DETAILED DESCRIPTION:
Children with spastic cerebral palsy often walk with insufficient ankle dorsiflexion in the swing phase or with eversion of the foot. A pathological gait, known as drop-foot gait, can be the result and this has 2 major complications: foot-slap during loading response and toe-drag during swing. This is partly caused by weakness of the anterior tibial muscle and partly due to co-contraction of both the fibular- and anterior tibial muscle. In time, the disorder appears to be progressive due to atrophy and contractures of the muscle and increasing bodyweight. For classification of gait, the Winters scale can be used, where unilateral CP with dropfoot is classified as type I.

In daily life these problems cause limited walking distance and frequent falls. This can lead to restrictions in participating in daily activities at school and in leisure. The current guideline for spastic cerebral palsy describes the following therapies: 1) conservative therapy, which includes physiotherapy, orthopaedic shoes and orthoses. 2) systemically and locally applied drugs suppressing spasticity. 3) surgical interventions, e.g. tenotomy, transposition and osteotomy. In each intervention, there is the risk of side effects, such as sedation with oral medications, pressure sores and atrophy in a static orthosis, temporary effect in a Botulinum toxin A treatment and surgical complications due to a result of the surgery, and on the other hand as a result of the execution.

Functional electrical stimulation (FES) may be an effective alternative treatment for children with spastic CP and a drop foot. By stimulating the fibular nerve or the anterior tibial muscle directly during the swing phase, dorsiflexion of the foot is stimulated. In contrast to bracing, FES does not restrict motion, but does produce muscle contraction, and thus has the potential to increase strength and motor control through repetitive neural stimulation over time.

In a systematic review the investigators found that FES immediately improves ankle dorsal flexion and falls. In addition, longer sustained effects of FES on ankle dorsal flexion and falls are found. However, it should be noted only two study studies (4 articles) were of level II class evidence (small RCT) and all other studies used a single subject design. Until now, the use of FES in CP is limited and no data exist about the effects on walking distance (activity level) and participation level.

The overall objective of this study is to conduct a randomised cross-over intervention trial in children with unilateral spastic CP with 12 weeks of FES for every participant and 18 weeks of conventional therapy. The effectiveness of FES will be examined at participation leven, using individual goal attainment. With every individual a goal at walking distance will be set, next to possible other goals. Next to that, results will be measured at the activity and functional level: the effect at gait kinematics (such as ankle dorsiflexion and balance), walking distance, falls, spasticity and muscle force. The type of brain damage of the patients is also taken in to account. An addition al goal is to investigate the cost effectiveness of FES, which, in case of a positive effect, may support allowance by insurance companies.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral foot drop of central origin, particularly the absence of initial heel contact
* Participants are currently treated with ankle-foot orthoses or (adapted) shoes to wear on a daily basis
* Participants ambulate independently, and thus classified as Gross Motor Function Classification System (GMFCS) levels I or II and have a gait type 1 according to Winters et al (4).
* Participants are able to walk for at least 15 minutes
* Confirmed cerebral abnormality with MRI (showing medial infarction, maldevelopment of the brain, or porencephaly).
* Participants are aged 4-18 years at time of inclusion

Exclusion Criteria:

* Plantarflexion ankle contracture of more than 5 degrees plantarflexion with the knee extended
* Botulinum toxin A injection to the plantar or dorsiflexor muscle groups within the 6 months before the study
* Orthopaedic surgery to the legs in the previous year
* Uncontrolled epilepsy with daily seizures

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in goal attainment scale (GAS) | Setting of goal(s) at start, assessment at every end of a phase: week 12, 18 and 30.
  Goal attainment scale: definition of an individual goal at start, followed by a 6- point numeric scale indicating to what extent the goal is (score 0 till +2) or is not (-3 indicating detoriation till -1) reached.

SECONDARY OUTCOMES:
Change in participation | assessment at start and every end of a phase: week 12, 18 and 30.
  as measured in the Cerebral Palsy Quality of Life Questionnaire (see reference).
Change in walking distance | assessment at start and every end of a phase: week 12, 18 and 30.
  Measured by the 6 minute walking test and the functional mobility scale (3 items, 6-point rating scale).
Change in physical activity | assessment at start and end of a phase (except for the wash-out phase): week 12 and 30.
  measured by activity monitor
Change in frequency of falling | assessment at every end of a phase: week 12, 18 and 30.
  measured by a questionnaire
Change in stability during walking | assessment at start and every end of a phase: week 12, 18 and 30.
  measured by variation of center of mass and margins of stability assessed during 3D gait analysis
Change in ankle dorsiflexion angle | assessment at start and every end of a phase: week 12, 18 and 30.
  measured in degrees during gait analysis during 3D gait analysis
Change in calf muscle activation | assessment at start and every end of a phase: week 12, 18 and 30.
  Assessed by spasticity measurement and electromyography (EMG) during 3D gait analysis
Change in ankle plantarflexion strength during walking | assessment at start and every end of a phase: week 12, 18 and 30.
  Calculated by net push off moments during 3D gait analysis
Change in ankle dorsiflexion and plantarflexion strength | assessment at start and every end of a phase: week 12, 18 and 30.
  measured in Newton by handheld dynamometer
Change in feelings about donning and doffing | assessment at start and every end of a phase: week 12, 18 and 30.
  measured by a questionnaire
Change in patient satisfaction | assessment at start and every end of a phase: week 12, 18 and 30.
  measured by a visual analogue scale with smileys (0 = unsatisfied, 6 = perfectly satisfied).
The compliance and acceptability of FES | the FES devices measures this automatically during wearing; so this will happen during the 12 weeks of FES therapy
  derived from delivered stimulations and hours of wear time in the log file
Type of brain lesion in relation to FES success | Assessment and analysis of available imaging will be done after completion of the study by the patient, so after week 30, up to week 50 to collect a batch of finished patients. No imaging will be performed because of the study.
  Derived from available brain imaging
Cost-effectiveness of FES | analysis after study completion, week 30, using the EQ-5D-Y results.
  compared to conventional therapy
Change in health | assessment at every end of a phase: week 12, 18 and 30.
  EQ-5D-Y Questionnaire, youth version

CONTACTS AND LOCATIONS:
Overall Officials: R.J. Vermeulen, prof M.D., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
With publishing our results, an additional data file will be available containing the original individual data (anonymized) in order to make meta-analysis possible.
Supporting Information: CSR
Time Frame: In the years 2020 and 2021.
Access Criteria: not yet known.

REFERENCES:
- [Background] Moll I, Vles JSH, Soudant DLHM, Witlox AMA, Staal HM, Speth LAWM, Janssen-Potten YJM, Coenen M, Koudijs SM, Vermeulen RJ. Functional electrical stimulation of the ankle dorsiflexors during walking in spastic cerebral palsy: a systematic review. Dev Med Child Neurol. 2017 Dec;59(12):1230-1236. doi: 10.1111/dmcn.13501. Epub 2017 Aug 17. PMID 28815571
- [Background] Waters E, Davis E, Mackinnon A, Boyd R, Graham HK, Kai Lo S, Wolfe R, Stevenson R, Bjornson K, Blair E, Hoare P, Ravens-Sieberer U, Reddihough D. Psychometric properties of the quality of life questionnaire for children with CP. Dev Med Child Neurol. 2007 Jan;49(1):49-55. doi: 10.1017/s0012162207000126.x. PMID 17209977
- [Derived] Moll I, Marcellis RGJ, Coenen MLP, Fleuren SM, Willems PJB, Speth LAWM, Witlox MA, Meijer K, Vermeulen RJ. A randomized crossover study of functional electrical stimulation during walking in spastic cerebral palsy: the FES on participation (FESPa) trial. BMC Pediatr. 2022 Jan 13;22(1):37. doi: 10.1186/s12887-021-03037-9. PMID 35027013
- See also: Pubmed link to the review — https://www.ncbi.nlm.nih.gov/pubmed/28815571